CLINICAL TRIAL: NCT01651468
Title: Phase 1 Study of the Nutraceutical "Hemofix" Safety and Effect on the Coagulation System
Brief Title: The Effect of the Nutraceutical "Hemofix" on the Coagulation System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The collaborator lost interest in a clinical study.
Sponsor: Hadassah Medical Organization (Other)
Collaborators: HEMOFIX (Unknown); Yocheved Grossman (Unknown); Idan Grossman (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HEMOFIX- HMO-CTIL
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-02

CONDITIONS: Von Willebrand Disease; Menorrhagia
Keywords: mild bleeding disorder
MeSH Terms: conditions — von Willebrand Diseases; Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HEMOFIX (Experimental): 3 grams a day
  Interventions: Dietary Supplement: HEMOFIX

INTERVENTIONS:
Dietary Supplement: HEMOFIX — unique complex herbal mixture

SUMMARY:
Hemofix is a herbal formula based on traditional Jewish and far eastern medicine created to assist in wound healing and bleeding arrest. It contains herbs such as Red Clover, Liquorice, Raspberry, Ginger and more. The present study will evaluate the formula on the coagulation system.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers and volunteers with a mild bleeding disorder

Exclusion Criteria:

* people with thrombophilic and cardiovascular complications,
* people who are treated with anti-coagulants,
* women taking birth control pills
* people with a history hypercoagulability

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2020-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
bleeding and blood test results | one year

CONTACTS AND LOCATIONS:
Overall Officials: David Varon, Prof, Principal Investigator — HMO
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel